CLINICAL TRIAL: NCT05265195
Title: PeriviAble DeLiveries: ALIgning PArental aNd PhysiCian PrioritiEs (ALLIANCE)
Acronym: ALLIANCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B01416
Record Dates: First submitted 2022-02-01; First posted 2022-03-03 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Periviable Infants; Extreme Prematurity; Communication
Keywords: Periviable Infant; Extreme Prematurity; Delivery Room Management; Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Semi-structured Interviews: Interviews will be conducted with parents and clinicians regarding their experiences of periviable counselling conversations. The interviews aim to identify key priorities and topic themes for the pre-delivery conversation for both parents and the clinicians, as these are hypothesised to differ between the groups.
  * Thematic analysis of transcribed semi-structured interviews with 20 parents and 20 clinicians.
  * The recruited parents will encompass a mixture of parent experiences: those with a surviving periviable child, parents whose baby died in delivery room and parents whose baby died in the neonatal unit.
  Interventions: Other: Mixed Methods study
- National evaluation of current periviable management practices across the UK.: Review of periviable deliveries and antenatal management practices in the United Kingdom for infants where the decision is for active care at delivery.
  Interventions: Other: Mixed Methods study
- Recording and thematic analysis of periviable decision-making conversations: * Recruiting parents who have presented in periviable labour to Manchester Foundation Trust sites.
  * Aiming to audio record 20 conversations discussing management options and potential outcomes between healthcare professionals and parents.
  * Thematic analysis will be undertake to determine key topics and priorities for parents and clinicians (these may well differ), time taken to discuss each topic, order topics presented, management options offered or requested, and discussion of comfort care.
  Interventions: Other: Mixed Methods study
- Comparison of recorded and simulated periviable decision-making conversations: * Recruit 20 senior clinicians from mixture of obstetric and neonatal specialities.
  * Clinician will participate in a standardised simulated discussion with two parents (played by actors) who have presented in periviable labour.
  * Simulated conversations will be audio recorded and transcribed.
  * Analysis will be performed for structure and topics included in this simulated conversation. Comparison will be undertaken comparing the conversational architecture of the simulated conversations with the recorded real conversations (recorded in the above phase of this study).
  Interventions: Other: Mixed Methods study
- Focus Groups with parents and clinicians: * Parent focus groups to consolidate and stratify key priority themes for periviable counselling and development of parent resources.
  * Clinician focus groups to discuss experiences with training in this area and preferences for future training methods/resources.
  * Parents will be recruited from parental advisory groups and local baby groups.
  * Aiming to run 5x focus groups with maximum 8 participants in each group.
  Interventions: Other: Mixed Methods study
- Parental survey of long-term outcomes: * Survey will be distributed to all parents of surviving periviable deliveries at St Mary's Manchester over the last 2 - 10 years.
  * Parents will be asked to complete the survey at home giving their views on their child's strengths, difficulties, development and social interactions.
  * The survey also asks parents for their views on what they remember they were told before they delivered and, in light of their experiences, what would they recommend clinicians include in pre-delivery periviable conversations with future parents.
  * The survey will be sent to all eligible parents, which equates to 220 surviving infants. All returned surveys will be analysed.
  Interventions: Other: Mixed Methods study

INTERVENTIONS:
Other: Mixed Methods study — Mixed Methods study

SUMMARY:
Background:

There is significant variation in how clinicians currently present information to parents in periviable labour. Whilst each conversation with an individual set of parents will vary, the current level of variation is extreme. In collaborative discussions with the neonatal parental advisory group whilst designing this project, parents reported numerous experiences of significant variation in practice between clinicians in relation to periviable delivery management. There is a pressing issue of injustice here as the hospital or clinician the parent presents to in labour should not restrict their access to information and options for management at delivery.

Parents should be empowered and engaged in making an individualised decision for their infant. However, this is not possible if information is not accurately presented to them. There is a gap in knowledge about what information is vital to include in periviable decision-making conversations between parents and healthcare professionals. This study aims to address this important gap in knowledge.

Research Question: How can information sharing and decision-making conversations between healthcare professionals and parents prior to periviable birth be improved?

Research Aims:

1. To gain understanding of current UK-wide antenatal optimisation practices for infants born at periviable gestations.
2. To establish an evidence-based conversational structure for pre-delivery periviable decision-making discussions, and a prioritised set of key discussion topics derived from parental consensus and clinician input.
3. To develop a set of parent and clinician derived recommendations to improve pre-delivery periviable decision-making conversations.

Methodology:

The study would progress along the following structure:

1. Literature Review of literature related to how and what information is presented to parents facing periviable labour by healthcare professionals.
2. Semi-structured interviews with clinicians and parents. The aim will be to determine an evidence-based set of priorities for each group and identify the differences in priorities and barriers that exist in communication between parents and clinicians.
3. National Evaluation of current periviable management practices across the UK. This will benchmark and expose variation in current practice.
4. Analysis of pre-delivery periviable conversations.
5. Focus groups with parents and clinicians to consolidate and stratify key priority themes for periviable decision-making conversations and assess acceptability of developing parent-centred periviable delivery resources.
6. Parent survey of parent-assessed long-term outcomes for periviable delivery survivors.

Impact and Dissemination:

This study will investigate the key topic areas and conversational structure of pre-delivery periviable decision-making conversations, aiming to provide evidence-based recommendations for improvement.

DETAILED DESCRIPTION:
Research Aims:

1. To gain understanding of current UK-wide antenatal optimisation practices for infants born at periviable gestations.
2. To establish an evidence-based conversational structure for pre-delivery periviable decision-making discussions, and a prioritised set of key discussion topics derived from parental consensus and clinician input.
3. To develop a set of parent and clinician derived recommendations to improve pre-delivery periviable decision-making conversations.

Research Objectives:

1. To benchmark current UK-wide antenatal optimisation intervention rates for periviable infants where active care has been deemed appropriate.
2. To record and perform thematic analysis of periviable decision-making conversations between parents and healthcare professionals.
3. To determine, then consolidate and stratify, key priority themes for periviable decision-making conversations using parent and clinician derived recommendations and avenues for dissemination.

Research Plan

1. Literature Review: Meta-synthesis of literature related to current pre-delivery periviable decision-making conversations and frameworks.
2. Semi-structured interviews:

   Aim: This study phase will determine an evidence-based set of priorities for each group and identify the differences in priorities and barriers that exist in communication between parents and clinicians. Semi-structured interviews will be conducted with 20 parents who have delivered a periviable baby and have experienced a range of outcomes after birth. There will also be interviews with 20 clinicians (equal split between obstetricians and neonatologists). Thematic analysis of the transcribed interviews will be performed to determine similarities and differences in parent and clinician experiences and priorities during pre-delivery periviable decision-making conversations.
3. National evaluation of current periviable management practices across the UK. Aim: This study phase will benchmark current periviable practices across the UK, evaluating the extent to which antenatal optimisation interventions (such as antenatal steroids) are utilised for periviable infants where active care was instigated after birth.
4. Recording and thematic analysis of periviable decision-making conversations. Aim: This study phase would involve recording real pre-delivery periviable decision-making conversations between clinicians and parents and analysing these for topics discussed, relative time spent on each topic and which management options at delivery were offered. Parents would be invited to participate in a follow-up interview 6 months later to evaluate if the pre-delivery conversation prepared them for the events that followed over their neonatal journey. This would aid evaluation of which conversations were helpful to parents and the structure of those helpful conversations could be used to inform better practice in the future.
5. Parent focus groups to consolidate and stratify key priority themes for periviable decision-making conversation and development of parent resources.

   Aim: This study phase will produce an evidence-based and parent-derived consensus of essential and desirable topic themes for inclusion in pre-delivery periviable decision-making conversations. These defined topic areas will provide a basis for future development of healthcare professional training curricula and the development of a parent information resource about periviable birth.
6. Parent survey of parent-assessed long-term outcomes for periviable delivery survivors.

Outcome:

This study will result in a set of evidence-based, prioritised topics for inclusion in periviable discussions between healthcare professional and parent. The study will also conclude with a set of recommendations for how to improve periviable discussion practices. The study results can be used as an evidence-basis to inform policy around periviable birth discussions and to develop clinician education curricula focused on translating the study results into improved everyday clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at periviable gestation. For this study periviability is defined as 22+0 - 24+6 weeks gestation.

Exclusion Criteria:

* Infants <22+0 or >24+6 weeks gestation.

Specific inclusion and exclusion criteria apply to each phase of the study.

Ages: 22 Weeks to 24 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will recruit a mixture of participants at various stages of the study:
  * Parents who have experienced a periviable labour,
  * Clinicians (Obstetricians, Midwives and Neonatologists) with experience of managing periviable deliveries.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Measures of current periviable delivery management: content of topics discussed in pre-delivery conversations and national rates of antenatal steroid and magnesium sulphate administration and place of birth. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Peterson, MBChB, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available to share. The study team are happy to share sections of anonymised transcripts from the study in the publication. However, no IPD will be available.